CLINICAL TRIAL: NCT05916833
Title: Comparison of Hypopressive Breathing and Noble Technique on Diastasis Recti Abdominis in Postpartum Women.
Brief Title: Comparison of Hypopressive Breathing and Noble Technique on DRA in Postpartum Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01536 Saima Awan
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Diastasis Recti Abdominis
Keywords: hypopressive; noble technique; DRA; postpartum women

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypopressive breathing technique (Experimental): These exercises involved "sucking in the abdomen" and opening the ribs by engaging the accessory inspiratory muscles, such as the serratus anterior, external intercostalis, scalenes, and sternocleidomastoid, while maintaining the glottis closed, a process known as "diaphragmatic suction.
  Interventions: Other: hypopressive breathing
- noble technique (Experimental): The Noble technique is (partially sitting up while manually flexing the rectus Abdominis muscles.
  Interventions: Other: noble technique

INTERVENTIONS:
Other: hypopressive breathing — Hot pack for 10min.Hypopressive breathing in sitting, lying and standing position. Hypopressive breathing 2 times/weekly, 5sec hold, 2-3reps, 1-2sets for 12 weeks. Session will be weekly progress.
  Arms: hypopressive breathing technique
Other: noble technique — Hot pack for 10min. Noble technique in relaxed supine position 2time/weekly, 3-5sec hold, 10-15reps, 2-3sets for 12 weeks. Session will be weekly progress.
  Arms: noble technique

SUMMARY:
The aim of study is to compare the effect of Hypopressive breathing and noble technique on width of Diastasis Recti Abdominis, lumbopelvic pain and maternal functioning in postpartum women.

DETAILED DESCRIPTION:
Candido shows that Caesarean section increased the likelihood of experiencing an increase in the inter-rectus distance during the postpartum period. Diastasis recti abdominis (DRA) is a common condition in postpartum women that can cause abdominal muscle separation. However, there is a lack of direct comparison between these two techniques. This study aims to compare the effectiveness of the hypopressive breathing and the Noble Technique in improving DRA in postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Multiparous women
* History of Cesarean section and vaginal delivery
* > 12 weeks postpartum
* Measurement is 2cm or more then 2cm of DRA is included by using finger width palpation and Nylon digital caliper
* Lumbopelvic pain (NPRS 3 to 8)

Exclusion Criteria:

* Exclude women who need surgical correction for DRA
* Pelvic organ prolapse
* Para umbilical hernia
* Malignancy
* Bone tuberculosis
* Fibromyalgia

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2023-02-04 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Modified OSWESTRY Low Back pain Index (ODI) | 12 weeks
  The Oswestry Low Back Pain Disability Index is a 10-point patient-reported outcome questionnaire that was first published in 1980. It is regarded as the "gold standard" for assessing quality of life (QoL) impairment and disability in persons with low back pain
IFSAC (Inventory of Functional Status After Childbirth) | 12 weeks
  The IFSAC consists of five subscales and 36 items, that is, infant care (6 items), personal care (8items), household activities (12 items), social and community activities (6 items), and occupational activities (4 items). The questionnaires are rated on a 4-point Likert scale and mean scores were calculated with one point being the lowest and four points being the highest scores possible.
Numeric Pain Rating Scale (NPRS): | 1 day
  The numeric pain rating scale (NPRS), a scoring system that quantifies pain on a scale from 0 (no pain) to 10 (worst possible agony), was used to determine the pain score.

CONTACTS AND LOCATIONS:
Overall Officials: summra andleeb, MS(OMPT), Principal Investigator — riphah internation university
Locations (1):
- Maryam's Clinic, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Axer H, Keyserlingk DG, Prescher A. Collagen fibers in linea alba and rectus sheaths. I. General scheme and morphological aspects. J Surg Res. 2001 Mar;96(1):127-34. doi: 10.1006/jsre.2000.6070. PMID 11181006
- [Background] Coldron Y, Stokes MJ, Newham DJ, Cook K. Postpartum characteristics of rectus abdominis on ultrasound imaging. Man Ther. 2008 May;13(2):112-21. doi: 10.1016/j.math.2006.10.001. Epub 2007 Jan 5. PMID 17208034
- [Background] Gilleard WL, Brown JM. Structure and function of the abdominal muscles in primigravid subjects during pregnancy and the immediate postbirth period. Phys Ther. 1996 Jul;76(7):750-62. doi: 10.1093/ptj/76.7.750. PMID 8677279
- [Background] 4. Gómez FR, Senín-Camargo FJ, Cancela-Cores Á, Patiño-Núñez S, Carballo-Costa L. C0083 Effect of a hipopressive abdominal exercise program on inter-rectus abdominis muscles distance in postpartum.
- [Background] Sperstad JB, Tennfjord MK, Hilde G, Ellstrom-Engh M, Bo K. Diastasis recti abdominis during pregnancy and 12 months after childbirth: prevalence, risk factors and report of lumbopelvic pain. Br J Sports Med. 2016 Sep;50(17):1092-6. doi: 10.1136/bjsports-2016-096065. Epub 2016 Jun 20. PMID 27324871
- [Background] Boissonnault JS, Blaschak MJ. Incidence of diastasis recti abdominis during the childbearing year. Phys Ther. 1988 Jul;68(7):1082-6. doi: 10.1093/ptj/68.7.1082. PMID 2968609
- [Background] Michalska A, Rokita W, Wolder D, Pogorzelska J, Kaczmarczyk K. Diastasis recti abdominis - a review of treatment methods. Ginekol Pol. 2018;89(2):97-101. doi: 10.5603/GP.a2018.0016. PMID 29512814
- [Background] Logsdon MC, Wisner KL, Pinto-Foltz MD. The impact of postpartum depression on mothering. J Obstet Gynecol Neonatal Nurs. 2006 Sep-Oct;35(5):652-8. doi: 10.1111/j.1552-6909.2006.00087.x. PMID 16958723
- [Background] Gjerdingen DK, Center BA. First-time parents' prenatal to postpartum changes in health, and the relation of postpartum health to work and partner characteristics. J Am Board Fam Pract. 2003 Jul-Aug;16(4):304-11. doi: 10.3122/jabfm.16.4.304. PMID 12949031
- [Background] Eriksson Crommert M, Petrov Fieril K, Gustavsson C. Women's experiences of living with increased inter-recti distance after childbirth: an interview study. BMC Womens Health. 2020 Nov 23;20(1):260. doi: 10.1186/s12905-020-01123-1. PMID 33228602
- [Background] Arranz-Martin B, Navarro-Brazalez B, Sanchez-Sanchez B, McLean L, Carazo-Diaz C, Torres-Lacomba M. The Impact of Hypopressive Abdominal Exercise on Linea Alba Morphology in Women Who Are Postpartum: A Short-Term Cross-Sectional Study. Phys Ther. 2022 Aug 4;102(8):pzac086. doi: 10.1093/ptj/pzac086. PMID 35908286
- [Background] Radhakrishnan M, Ramamurthy K. Efficacy and Challenges in the Treatment of Diastasis Recti Abdominis-A Scoping Review on the Current Trends and Future Perspectives. Diagnostics (Basel). 2022 Aug 24;12(9):2044. doi: 10.3390/diagnostics12092044. PMID 36140446
- [Background] Lee D, Hodges PW. Behavior of the Linea Alba During a Curl-up Task in Diastasis Rectus Abdominis: An Observational Study. J Orthop Sports Phys Ther. 2016 Jul;46(7):580-9. doi: 10.2519/jospt.2016.6536. PMID 27363572
- [Background] Davenport MH, Marchand AA, Mottola MF, Poitras VJ, Gray CE, Jaramillo Garcia A, Barrowman N, Sobierajski F, James M, Meah VL, Skow RJ, Riske L, Nuspl M, Nagpal TS, Courbalay A, Slater LG, Adamo KB, Davies GA, Barakat R, Ruchat SM. Exercise for the prevention and treatment of low back, pelvic girdle and lumbopelvic pain during pregnancy: a systematic review and meta-analysis. Br J Sports Med. 2019 Jan;53(2):90-98. doi: 10.1136/bjsports-2018-099400. Epub 2018 Oct 18. PMID 30337344
- [Background] van de Water AT, Benjamin DR. Measurement methods to assess diastasis of the rectus abdominis muscle (DRAM): A systematic review of their measurement properties and meta-analytic reliability generalisation. Man Ther. 2016 Feb;21:41-53. doi: 10.1016/j.math.2015.09.013. Epub 2015 Oct 3. PMID 26474542
- [Background] Mousavi SJ, Parnianpour M, Mehdian H, Montazeri A, Mobini B. The Oswestry Disability Index, the Roland-Morris Disability Questionnaire, and the Quebec Back Pain Disability Scale: translation and validation studies of the Iranian versions. Spine (Phila Pa 1976). 2006 Jun 15;31(14):E454-9. doi: 10.1097/01.brs.0000222141.61424.f7. PMID 16778675
- [Background] Noor NM, Aziz AA, Mostapa MR, Awang Z. Validation of the Malay version of the Inventory of Functional Status after Childbirth questionnaire. Biomed Res Int. 2015;2015:972728. doi: 10.1155/2015/972728. Epub 2015 Jan 15. PMID 25667932
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Navarro-Brazalez B, Prieto-Gomez V, Prieto-Merino D, Sanchez-Sanchez B, McLean L, Torres-Lacomba M. Effectiveness of Hypopressive Exercises in Women with Pelvic Floor Dysfunction: A Randomised Controlled Trial. J Clin Med. 2020 Apr 17;9(4):1149. doi: 10.3390/jcm9041149. PMID 32316686